CLINICAL TRIAL: NCT01560598
Title: Adipokines and the Risk of Reflux Esophagitis : Prospective Case-control Study
Brief Title: Adipokines and the Risk of Reflux Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Donghee Kim, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: gerdadipokine
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Visceral Obesity; Reflux Esophagitis
Keywords: GERD; reflux esophagitis; adipokine; especially; endoscopically proven
MeSH Terms: conditions — Obesity, Abdominal; Esophagitis, Peptic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Reflux esophagitis: those with endoscopically proven reflux esophagitis
- Normal: those with normal GFS finding (without definite mucosal break at Z-line)

SUMMARY:
We aimed to risk faoctors for GERD and association between visceral obesity, plasma adipoline(leptin, adiponectin, IL-6, TNF-α)and development of reflux esophagitis in healthy Koreans.

ELIGIBILITY:
Inclusion Criteria:

* endoscopically proven reflux esophagitis

Exclusion Criteria:

* those with esophageal hiatal hernia, current PPI medication, upper GI operation history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults who visit healthcare system for routine checkup
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Difference in serum adipokine levels between case and control groups | 2 month lager (after sampling)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Healthcare System Gangnam Center, Seoul, South Korea